CLINICAL TRIAL: NCT05796752
Title: Single-Group Crossover Trial Comparing Behavioral Treatment to Memantine in Body Focused Repetitive Behaviors
Brief Title: Behavioral Treatment and Memantine in Body Focused Repetitive Behaviors
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB23-0033
Record Dates: First submitted 2023-03-22; First posted 2023-04-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-09

CONDITIONS: Skin-Picking; Trichotillomania (Hair-Pulling Disorder)
MeSH Terms: conditions — Excoriation Disorder; Trichotillomania | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Memantine and Behavioral Therapy (Experimental): All subjects will receive 8-weeks of memantine treatment (10mg po qday for the first two weeks, then 20 mg po qday for the remaining six weeks). After the 8-weeks of memantine treatment, the dose will be discontinued. Then, after a 4-week washout period, all subjects will receive 8-weeks of ComB therapy. Therapy will be once a week for 30 minutes. After the 8-weeks of ComB treatment, the therapy will be discontinued.
  Interventions: Drug: Memantine; Behavioral: ComB Behavioral Therapy

INTERVENTIONS:
Drug: Memantine — Cognition-enhancing medication
  Other Names: Namenda
Behavioral: ComB Behavioral Therapy — Therapy for BFRBs

SUMMARY:
The goal of the proposed study is to compare the efficacy of behavioral treatment (BT) to memantine, a psychopharmacological agent, for BFRBs. 28 subjects with trichotillomania (TTM) or skin picking disorder (SPD) will receive 8 weeks of memantine treatment, followed by 8 weeks of comprehensive behavioral therapy (ComB) treatment. The hypothesis to be tested is that behavioral therapy will be associated with superior clinical outcomes as compared to memantine. A second hypothesis is that both memantine and behavioral therapy will demonstrate improvement from baseline to the respective posttreatment assessment.

DETAILED DESCRIPTION:
Hair pulling disorder (i.e., trichotillomania, TTM) and skin picking disorder (SPD) are often categorized under the umbrella term of BFRB disorders. These repetitive, intentionally performed behaviors often cause noticeable cosmetic issues and may result in clinically significant distress or functional impairment.

Behavioral therapy (BT) is generally regarded as the first-line treatment for BFRBs. One type of BT is comprehensive behavioral treatment (ComB), a treatment that emphasizes habit reversal training and various techniques that target specific BFRB triggers (e.g., sensory cues, such as pressure on the scalp; environmental cues, such as bright lights and mirrors), including emotion dysregulation. The ComB protocol was methodically developed based on expert consensus and demonstrated promising results in one single case design study and a randomized controlled trial comparing it to a minimal attention control condition.

Research has also found benefit of pharmacological agents in the treatment of BFRBs. Most recently, a randomized controlled trial of memantine vs. placebo found statistically significant improvements in disorder severity and life functioning in the memantine group as compared to the placebo group.

Although there are emerging behavioral and psychopharmacological interventions for BFRBs, the research is limited. Additionally, there are no studies comparing the efficacy of first-line behavioral treatments to promising medication interventions for this class of disorders. Given the serious personal consequences associated with trichotillomania and skin picking disorder, there is substantial need for additional research to clarify the best available treatments for BFRBs. Doing so would facilitate future research and the development of refined treatment guidelines. Therefore, the current trial aims to compare the efficacy of behavioral therapy and memantine in adults with trichotillomania and skin picking disorder.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18+
* Current DSM-5 diagnosis of trichotillomania (TTM) or skin picking disorder (SPD)
* Ability to understand and sign the consent form
* Stable dose of medications for at least the past 3 months

Exclusion Criteria:

* Unstable medical illness based on history or clinically significant abnormalities on baseline physical examination
* Current pregnancy or lactation, or inadequate contraception in women of childbearing potential
* Subjects considered an immediate suicide risk based on the Columbia Suicide Severity rating Scale (C-SSRS)
* Past 12-month DSM-5 diagnosis of psychosis, bipolar disorder, mania, or a substance or alcohol use disorder
* Illegal substance use based on urine toxicology screening
* Previous treatment with memantine
* Previous trial of ComB or similar BT protocol (e,g., habit reversal training)
* Cognitive impairment that interferes with the capacity to understand and self-administer medication or provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
National Institutes of Mental Health Symptom Severity Scale (for trichotillomania or Skin Picking) (NIMH-TSS or NIMH-SPS) | The primary efficacy endpoints will be the change in these measures from baseline to week 8 in memantine treatment vs. ComB treatment.
  The primary efficacy measure will be the change in hair pulling or skin picking frequency and urges to pull hair or pick skin for the past week as indicated by change in total score on the NIMH Symptom Severity Scale (for Trichotillomania or Skin Picking). The primary endpoints will be used to examine differential improvements for memantine vs. BT. Total scores on the NIMH-TSS and NIMH-SPS range from 0-20, with higher scores representing greater severity of trichotillomania/skin picking.

SECONDARY OUTCOMES:
Clinical Global Impressions -- Improvement Scale (CGI-I) | 20 weeks
  A clinician-rated measure to assess global improvement in symptoms. The scale ranges from 1 (Very much improved) to 7 (Very much worse). The results will be dichotomized as improved (CGI-I score of 1 or 2) or not improved (CGI-I score of 3-7). The scale will be assessed at the end of the memantine treatment, at the end of the washout period, and at the end of the ComB therapy treatment.
Massachusetts General Hospital Hairpulling Scale (MGH-HPS) | 20 weeks
  Brief, self-report instrument for assessing repetitive hairpulling. Seven individual items, rated for severity from 0 to 4, assess urges to pull, actual pulling, perceived control, and associated distress. Total scores range from 0-28, with higher scores indicating greater severity of trichotillomania (TTM).The scale will be administered at screening, the end of the memantine treatment, at the end of the washout period, and at the end of the ComB therapy treatment.
Massachusetts General Hospital Hairpulling Scale -- Revised for Skin Picking | 20 weeks
  Brief, self-report instrument for assessing repetitive skin picking. Seven individual items, rated for severity from 0 to 4, assess urges to pick, actual picking, perceived control, and associated distress. Total scores range from 0-28, with higher scores indicating greater severity of skin picking disorder. The scale will be administered at screening, the end of the memantine treatment, at the end of the washout period, and at the end of the ComB therapy treatment.
Quality of Life Inventory | 20 weeks
  A self-report assessment of patient perceived quality of life. Quality of Life Inventory t-scores range from 1-77. Higher scores indicate a higher quality of life, whereas lower scores indicate a lower quality of life. The scale will be administered at screening, the end of the memantine treatment, at the end of the washout period, and at the end of the ComB therapy treatment.
Sheehan Disability Scale (SDS) | 20 weeks
  A self-report measure of functional impairment from TTM or SPD. SDS total scores range from 0-30. Higher scores indicate greater functional impairment. The scale will be administered at screening, the end of the memantine treatment, at the end of the washout period, and at the end of the ComB therapy treatment.
Hamilton Anxiety Rating Scale (HAM-A) | 20 weeks
  A clinician-administered assessment of anxiety. HAM-A total scores range from 0-56. Higher scores indicate higher levels of anxiety, with 0 being no symptoms of anxiety. The scale will be administered at screening, the end of the memantine treatment, at the end of the washout period, and at the end of the ComB therapy treatment.
Hamilton Depression Rating Scale (HAM-D) | 20 weeks
  A clinician-administered assessment of depression. HAM-D total scores range from 0-52. Higher scores indicate higher levels of depression, with 0 being no symptoms of depression. The scale will be administered at screening, the end of the memantine treatment, at the end of the washout period, and at the end of the ComB therapy treatment.
Barratt Impulsiveness Scale (BIS) | 20 weeks
  A self-report assessment of impulsivity. BIS total scores range from 30-120. Higher total scores indicate higher impulsiveness. The scale will be administered at screening, the end of the memantine treatment, at the end of the washout period, and at the end of the ComB therapy treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jon E Grant, MD, JD, MPH, Principal Investigator — University of Chicago; Gregory Chasson, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Grant JE, Chamberlain SR. Trichotillomania. Am J Psychiatry. 2016 Sep 1;173(9):868-74. doi: 10.1176/appi.ajp.2016.15111432. PMID 27581696
- [Background] Woods DW, Flessner CA, Franklin ME, Keuthen NJ, Goodwin RD, Stein DJ, Walther MR; Trichotillomania Learning Center-Scientific Advisory Board. The Trichotillomania Impact Project (TIP): exploring phenomenology, functional impairment, and treatment utilization. J Clin Psychiatry. 2006 Dec;67(12):1877-88. doi: 10.4088/jcp.v67n1207. PMID 17194265
- [Background] Grant JE, Odlaug BL, Chamberlain SR, Keuthen NJ, Lochner C, Stein DJ. Skin picking disorder. Am J Psychiatry. 2012 Nov;169(11):1143-9. doi: 10.1176/appi.ajp.2012.12040508. PMID 23128921
- [Background] Farhat LC, Olfson E, Nasir M, Levine JLS, Li F, Miguel EC, Bloch MH. Pharmacological and behavioral treatment for trichotillomania: An updated systematic review with meta-analysis. Depress Anxiety. 2020 Aug;37(8):715-727. doi: 10.1002/da.23028. Epub 2020 May 10. PMID 32390221
- [Background] Falkenstein MJ, Mouton-Odum S, Mansueto CS, Golomb RG, Haaga DA. Comprehensive Behavioral Treatment of Trichotillomania: A Treatment Development Study. Behav Modif. 2016 May;40(3):414-38. doi: 10.1177/0145445515616369. Epub 2015 Dec 7. PMID 26643276
- [Background] Bottesi G, Ouimet AJ, Cerea S, Granziol U, Carraro E, Sica C, Ghisi M. Comprehensive Behavioral Therapy of Trichotillomania: A Multiple-Baseline Single-Case Experimental Design. Front Psychol. 2020 Jun 10;11:1210. doi: 10.3389/fpsyg.2020.01210. eCollection 2020. PMID 32587552
- [Background] Carlson EJ, Malloy EJ, Brauer L, Golomb RG, Grant JE, Mansueto CS, Haaga DAF. Comprehensive Behavioral (ComB) Treatment of Trichotillomania: A Randomized Clinical Trial. Behav Ther. 2021 Nov;52(6):1543-1557. doi: 10.1016/j.beth.2021.05.007. Epub 2021 Jun 3. PMID 34656205
- [Background] Swedo SE, Leonard HL, Rapoport JL, Lenane MC, Goldberger EL, Cheslow DL. A double-blind comparison of clomipramine and desipramine in the treatment of trichotillomania (hair pulling). N Engl J Med. 1989 Aug 24;321(8):497-501. doi: 10.1056/NEJM198908243210803. PMID 2761586
- [Background] Keuthen NJ, O'Sullivan RL, Ricciardi JN, Shera D, Savage CR, Borgmann AS, Jenike MA, Baer L. The Massachusetts General Hospital (MGH) Hairpulling Scale: 1. development and factor analyses. Psychother Psychosom. 1995;64(3-4):141-5. doi: 10.1159/000289003. PMID 8657844
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] HAMILTON M. The assessment of anxiety states by rating. Br J Med Psychol. 1959;32(1):50-5. doi: 10.1111/j.2044-8341.1959.tb00467.x. No abstract available. PMID 13638508
- [Background] Patton JH, Stanford MS, Barratt ES. Factor structure of the Barratt impulsiveness scale. J Clin Psychol. 1995 Nov;51(6):768-74. doi: 10.1002/1097-4679(199511)51:63.0.co;2-1. PMID 8778124